CLINICAL TRIAL: NCT06621407
Title: Active 24 Hours Subperiostal vs. 24 Hours Passive Subdural Drainage Following Burr Hole Evacuation of Chronic Subdural Hematoma (the SUPERDURA Trial) - Protocol for a Nationwide Randomized Clinical Non-inferiority Trial
Brief Title: A National Study Examining the Most Effective Drainage Method After Burr Hole Evacuation of Chronic Subdural Hematoma
Acronym: SUPERDURA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University Hospital (Other)
Collaborators: Odense University Hospital (Other); Rigshospitalet, Denmark (Other); Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Carsten Reidies Bjarkam, Professor, Senior Consultant, Aalborg University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: N-20240009
Record Dates: First submitted 2024-09-19; First posted 2024-10-01 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Chronic Subdural Hematoma; Surgical Procedures, Operative; Recurrence; Mortality; Drainage; Drainage/Methods; Drainage Procedure
MeSH Terms: conditions — Hematoma, Subdural, Chronic; Recurrence

STUDY DESIGN:
Intervention Model Description: Randomized multicenter clinical non-inferiority trial encompassing all neurosurgical units in Denmark. All adult patients with symptomatic unilateral CSDH admitted to a Danish neurosurgical unit for single burr hole evacuation will be considered for inclusion. Before surgical hematoma evacuation patients will be randomized to 24 hours passive subdural drainage or 24 hours active subperiostal drainage, and the drain placed accordingly at the end of the hematoma evacuation procedure. The primary end point is a composite outcome of 90-day mortality, and recurrent CSDH on the same side as the primary operation requiring reoperation within the 90-day follow-up period.
Who Masked: Participant, Outcomes Assessor
Masking Description: Due to the inherent nature of the intervention blinding of the treating personnel is not possible. However, patients, the study statisticians, the 90-day outcome assessors, and the study steering group will be blinded to the allocation. Furthermore, statistical analyses and initial interpretation of the results will be performed using data with blinded treatment allocation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 24 hours active subperiostal drainage (Experimental): 24 hours active subperiostal drainage after single burr hole evacuation of a chronic subdural hematoma
  Interventions: Procedure: 24 hours active subperiostal drainage
- 24 hours passive subdural drainage (Experimental): 24 hours passive subdural drainage after single burr hole evacuation of a chronic subdural hematoma
  Interventions: Procedure: 24 hours passive subdural drainage

INTERVENTIONS:
Procedure: 24 hours active subperiostal drainage — 24 hours active subperiostal drainage after single burr hole evacuation of a chronic subdural hematoma
  Arms: 24 hours active subperiostal drainage
Procedure: 24 hours passive subdural drainage — 24 hours passive subdural drainage after single burr hole evacuation of a chronic subdural hematoma
  Arms: 24 hours passive subdural drainage

SUMMARY:
Chronic subdural hematoma (CSDH) is a common disease. The main treatment is neurosurgical evacuation and subsequent hematoma drainage. However, consensus on the optimal drain placement site, and whether the drainage should be active or passive, is lacking.

The aim of the current study is to test the hypothesis that 24 hours active subperiosteal drainage is non-inferior to 24 hours passive subdural drainage after single burr hole evacuation of a unilateral CSDH.

The study is a multicenter randomized non-inferiority trial encompassing all neurosurgical units in Denmark.

Adult patients with symptomatic CSDH admitted to a Danish neurosurgical unit for single burr hole evacuation will be screened for inclusion. Patients who are not able to give informed consent, and patients with recurrent CSDH, known cerebrospinal fluid abnormalities, and other known brain pathologies will be excluded. Patients with bilateral CSDH will be registered as one case and treated similarly on both sides.

Before surgical hematoma evacuation patients will be randomized to 24-hour passive subdural drainage or 24-hour active subperiosteal drainage.

The patients included and the two study statisticians will be blinded. The primary outcome is a composite outcome of 90-day mortality and symptomatic CSDH recurrence.

Secondary outcomes are 90-day simplified modified Rankin score (smRSq), and complications related to surgery or occurring during admission, including intracerebral hemorrhage due to misplaced drains, acute subdural hematoma, tension pneumocephalus, wound infection, drain seepage, subperiosteal hematoma, thromboembolic events, infections and seizures.

Sample size simulations of non-inferiority with a threshold of 7% increased relative risk show that a total of 354 participants will be required to demonstrate a relative risk reduction of recurrent CSDH and mortality of 30% for the cohort receiving active subperiosteal drainage given a stable power above 80% with an alpha of 5%. The study inclusion period is estimated to last 2 years.

Ethics approval for inclusion of competent patients has been obtained (N-20240009).

DETAILED DESCRIPTION:
The incidence of symptomatic chronic subdural hematoma (CSDH) is sharply on the rise due to an ageing population, and population risk factors such as alcohol misuse, falls, and use of anticoagulants and -platelets. The treatment of symptomatic CSDH is neurosurgical hematoma evacuation followed by drain placement to facilitate subsequent postoperative drainage. Accordingly, in many general neurosurgical departments this is the most common cranial procedure performed on a daily basis. However, no consensus exists on the actual surgical technique (hematoma evacuation by one burr hole, more burr holes or a larger cranial opening (craniotomy), hematoma irrigation method, drain placement site (subdural or subperiostal), and drainage method (time, active versus passive). This was also the case in Denmark where the actual CDSH evacuation technique differed vastly between departments and between neurosurgeons at the same department, although there only were four neurosurgical units in Denmark treating patients with symptomatic CSDH. Accordingly, in 2012 on the initiative of the four Danish neurosurgical departments the Danish Chronic Subdural Hematoma group (DACSUHS) was established in order to generate evidence based guidelines for the treatment of CSDH, standardize the treatment, and conduct national multicenter CSDH research. The first national CSDH treatment guideline was based on data collected retrospectively from 2010 to 2012, rigorous literature search, and a concluding Delphi process in the DACSUHS consortium, before it was finally published in 2018. It reflects the best available evidence regarding 10 aspects of CSDH management, including preoperative evaluation, surgical approach, postoperative mobilization, and use of postoperative head CT. Furthermore, it enabled the standardization of the CSDH treatment in all Danish departments by requiring the use of the same operative technique, drains, fixation technique for drains, and written patient information. The standardized CSDH approach enabled also the initiation of two larger prospective national multicenter trials evaluating the optimal postoperative drainage time in relation to CSDH recurrence rate and patient mortality. These above-mentioned process steps haves resulted in the current Danish CSDH treatment algorithm recommending evacuation of symptomatic CSDH by a single perforator made 13-mm burr hole above the maximum width of the hematoma followed by subdural temperate isotonic saline irrigation and subsequent placement of a subdural drain for 24 hours.

The subdural drain placement has, however, been much debated as drain placement through the skull burr hole in the subdural space in direct proximity to the brain may result in brain lesions, bleeding, seizures, and intracranial infections.

Therefore, burr hole craniostomy with subperiosteal drainage (also known as subgaleal drainage) has been suggested as an equally safe and effective treatment of CSDH due to less invasiveness and lower risk of drain inflicted brain parenchyma injury.

Neurosurgeons have generally been reluctant to use active (vacuum) drainage on subdural drains due to their proximity to the brain, whereas active drainage is more common active with subperiostal drainage has been more common. Although a direct comparison is lacking, it has been shown in a paper comparing three different Scandinavian centers using active subperiostal drainage, passive subdural drainage, and subdural drainage with continuously irrigation, that patients receiving passive drainage had the highest recurrence rate (20% vs. 11%) and on average a slightly higher complication rate (8.1% vs. 7.3%) and mortality rate (7.3% vs. 5.8%) compared to active subperiostal drainage which had a recurrence rate of 11.1% and a complication and mortality rate of 7.3% and 5.8%, respectively. Similarly, Post-hoc analysis of the cSDH-Drain and the TOSCAN studies have likewise revealed a higher recurrence rate (23.1% vs 14.1%) in patients receiving passive compared to active drainage.

Accordingly, as active subperiostal drainage might seem to be more safe and more efficient, the investigators find it justified to examine if 24 hours active subperiostal drainage is non-inferior to our current gold standard of 24 hours passive subdural drainage in a randomized clinical trial (the SuperDura trial).

The obtained results from the SuperDura trial will not only have major relevance for neurosurgical praxis as the investigators perform the first direct comparison between two commonly used drainage methods on a national level.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥ 18 years).
* Patients with symptomatic CSDH confirmed on brain CT- or magnetic resonance imaging (MRI), admitted to a Danish neurosurgical department for surgical treatment.
* Patients undergoing a single burr-hole evacuation.
* Informed written and oral consent is taken prior to surgery.

Exclusion Criteria:

* Patients who are mentally incapacitated
* Patients with known abnormalities in their cerebrospinal fluid (protein and glucose levels, cell count, and type)
* Patients with changes or abnormalities in their normal cerebrospinal fluid dynamics, e.g., obstructive hydrocephalus, normal pressure hydrocephalus, intracranial hypotension, and ventricular peritoneal shunt.
* Patients with additional/previously intracranial pathology that requires/has required neurosurgical treatment (e.g., brain tumor, vascular malformation, abscess).
* Patients with recurrent CSDH or with previous craniotomy or other transcranial surgery (for any reason)
* Patients unable to give consent prior to surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 354 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Composite outcome of 90-day mortality and recurrent CSDH on the same side as the primary operation requiring reoperation within the 90-day observation period | From enrollment to 90-days postsurgery
  The primary outcome measure is a composite outcome of 90-day mortality and recurrent CSDH on the same side as the primary operation requiring reoperation within the 90-day observation period. Recurrent CSDH is defined as a re-accumulation of the previously treated CSDH requiring ipsilateral or bilateral reoperation following symptom improvement after the first operation. For both unilateral and bilateral hematomas, recurrence will be considered as one reoperation.

SECONDARY OUTCOMES:
90-day simplified modified Rankin scale | 90 days after enrollment
  The scores on the simplified modified Rankin scale will be assessed with the use of the simplified mRS validated questionnaire, which will be completed over the telephone by the patients or next of kin at 90 (80-100) days after surgery. The results will be dichotomized and analyzed with 0-2 as favourable clinical outcome and 3-6 as unfavourable outcome.
90-day serious adverse events (SAE) | From time of surgery to 90-days postoperative
  Serious adverse events (SAE) necessitating new hospitalization in the 90 days postoperative period
Complications related to surgery | From enrollment to 90-days postsurgery
  Complications related to surgery encompasing intracerebral hemorrhage due to misplaced drains, acute subdural hematoma, tension pneumocephalus, wound infection, drain seepage, subperiostal hematoma, and seizures.
Postoperative adverse events during the admission | From enrollment to admission from hospital assessed up to 90-days postsurgery
  Postoperative adverse events during the admission emcompassing thromboembolic events and/or infections.
Length of hospitalization | From enrollment to admission from neurosurgical department, and from surgical CSDH evacuation to discarge to home or nursing facility, assessed up to 90-days postsurgery
  Length (days) of admission to neurosurgical department. Length (days) of hospitalization in total after surgical CSDH evacuation
Simplified mRSq as an ordinal outcome | 90-days postoperative
  Ordinal predentation of the 90-day simplified mRSq.
90-day mortality and registered cause of death. | From enrollment to 90-days postsurgery
  Mortality within 90 days of the performed surgery
  Registred cause of death
90-day recurrent symptomatic CSDH requiring ipsilateral or bilateral reoperation within 90 days. | From surgery to 90-day postsurgery
  Recurrent symptomatic CSDH requiring ipsilateral or bilateral reoperation within 90 days. For both unilateral and bilateral hematomas, recurrence will be considered as one reoperation.
Discharge destination | From enrollment to 90-days postsurgery
  Discharge destination after completed neurosurgical CSDH evacuation encompassing home, nursing home, other hospital department

OTHER OUTCOMES:
Use of antithrombotics | From admission to 90-days postoperative
  Use of antithrombotic (its preoperative time of cessation, and its postoperative time of restart). Related to the primary outcome.
Time to surgery | From adimission to time of surgery
  Time to surgery (split between median time of population) related to the primary outcome
Unilateral versus bilateral CSDH | From admission to 90 days postoperative
  Unilateral versus bilateral CSDH related to the primary outcome
Recurrence rate per hematoma side | From surgery to 90 days postoperative
  Symptomatic CSDH recurrence requiring operation counted pr hematoma side

CONTACTS AND LOCATIONS:
Overall Officials: Carsten R Bjarkam, MD, PhD, DMSc, Study Director — Department of Neurosurgery, Aalborg University Hospital, Denmark
Locations (4):
- Denmark (4):
  - Department of Neurosurgery, Aalborg University Hospital, Aalborg
  - Department of Neurosurgery, Aarhus University Hospital, Aarhus
  - Department of Neurosurgery, Copenhagen University Hospital Rigshospitalet, Copenhagen
  - Department of Neurosurgery, Odense University Hospital, Odense

IPD SHARING:
Plan to Share IPD: Yes
All collected data will be shared in annonymized form.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: From December 1st 2024 to November 30th 2032
Access Criteria: A written request to gain access to the datasets obtained during this study can be sent to the corresponding author, which will be discussed in the DACHSUS research team. If approved, the corresponding author will be responsible for providing access to research data requested by third parties, unless access to the data is restricted by a legal obligation (e.g., non-disclosure agreement), intellectual property protection, ethical approval requirements, ethical or security reasons, or other legitimate reasons.

REFERENCES:
- [Background] Hjortdal Gronhoj M, Jensen TSR, Miscov R, Sindby AK, Debrabant B, Hundsholt T, Bjarkam CR, Bergholt B, Fugleholm K, Poulsen FR; DACSUHS group. Optimal drainage time after evacuation of chronic subdural haematoma (DRAIN TIME 2): a multicentre, randomised, multiarm and multistage non-inferiority trial in Denmark. Lancet Neurol. 2024 Aug;23(8):787-796. doi: 10.1016/S1474-4422(24)00175-3. Epub 2024 Jun 12. PMID 38878790
- [Derived] Terkelsen JH, Miscov R, Jensen TSR, Schack A, Gronhoj MH, Korshoj AR, Haldrup M, Poulsen FR, Fugleholm K, Bjarkam CR, Olsen MH. Active subperiosteal vs. passive subdural 24-h drainage following single burr hole evacuation of chronic subdural hematoma: statistical analysis plan for the multicenter, randomized, non-inferiority clinical trial SUPERDURA. Trials. 2026 Jan 17. doi: 10.1186/s13063-026-09434-8. Online ahead of print. PMID 41546119